CLINICAL TRIAL: NCT04242043
Title: Feasibility Study for Improving the Relevance of Diagnostic Proposals for an Artificial Intelligence Software in the Elderly Population.
Acronym: Intel@Med-Fais
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0026 (Intel@Med-Faisa)
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2021-10

CONDITIONS: Artificial Intelligence; Geriatrics; Diagnostic Proposals Elderly
Keywords: Artificial Intelligence; Geriatrics; diagnostic proposals elderly

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AI
  Interventions: Diagnostic Test: intel@med-feasibility

INTERVENTIONS:
Diagnostic Test: intel@med-feasibility — Initial evaluation by the Nurse using the AI tool which enters into MEDVIR the patient's symptoms or functional complaints and comorbidities and is complemented by a telemedicine solution for data transmission to the remote tele-expert physician located in a regulatory center or health center. The remote doctor (a geriatrician from "Prevention Care for Elderly Unit (UPSAV) platform" of the Clinical Gerontology Division of the Limoges University Hospital) analyses the data collected by the Nurse and establishes a symptom severity criterion and a diagnosis with the help of the AI technology.
  Both the geriatrician and the NHs nurse are not aware of the proposals made by AI.
  The geriatrician can nevertheless initiate a visit to the resident's place of residence in order to verify the information necessary to establish the diagnosis and thus improve the relevance of the algorithm. For the resident, this study doesn't interfere with the usual care.

SUMMARY:
The ageing of the population is accompanied by the problem of chronic pathologies and sometimes heavy dependence, requiring admission to Nursing Homes (NHs). Approximately 660,000 people currently live in NHs in France. One out of 3 NHs does not have a coordinating doctor, even though the law requires it, and access to care in these NHs is very unequal nationally and especially in the Limousin and Dordogne regions. Some Hospices may find themselves in a situation where there is no coordinating doctor and difficult access to General Practitioners (GPs) visiting a large area.

This inequality of access to care results in a difference in care that can go as far as a loss of opportunity for residents who are immediately transferred to the emergency department (ED) with a risk of iatrogeny or delirium once in the ED or a risk of inappropriate hospitalization.

Residents are hospitalized:

* when the latter could have been avoided because the health care team, not knowing what attitude to adopt, prioritized hospitalization
* Late because the resident waited for the attending physician to come, which resulted in a worsening of symptoms.

The arrival of Artificial Intelligence (AI) is an opportunity to find new models of care organization that can mitigate medical desertification but also develop advanced practices in gerontology. For example, nurses will be able to intervene at a first level for early detection, better triage and early management of certain pathologies.

The "MEDVIR society" AI, developed by a French company, is a medical decision support system with Artificial Intelligence and offers pre-diagnosis based on the information collected (medical and surgical history, concomitant treatments and symptoms). MEDVIR is a diagnostic aid tool and does not replace the doctor who remains at the end of the chain, the final decision-maker.

Before research is conducted to integrate this technology into routine care, it is important to validate the diagnostic relevance of AI in the elderly, as it has been validated in the general population.

This pilot feasibility study will then enable us to methodologically dimension a future project to evaluate the efficiency of this new care system in the management of elderly patients in medical deserts in France.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 or over
* Patient living in one of the two NHs tests
* Patient with a functional complaint or abnormal symptoms involving the call of a physician
* Patient or his legal representative who has not expressed his opposition to the collection of his medical and personal data
* Patient affiliated to social security

Exclusion Criteria:

* End-of-life patient
* Patient with a clear vital emergency according to the physician
* Chronic aphasic patient

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Resident in nursing home presenting a health problem that requires the call of his/her attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-12-21 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
AI diagnostic proposals | 1 month
  Number of AI diagnostic proposals in adequacy with the medical diagnosis in the month of the study

SECONDARY OUTCOMES:
severity diagnoses | 1 month
  Number of severity diagnoses proposed by the AI solution versus medical diagnosis of the remote geriatrician over the month of the study
satisfaction survey | 1 month
  Analysis of the satisfaction survey filled in by the users (NHs nurses, participants, NHs Directors and geriatricians)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ehpad Des Bayles, Isle
  - Ehpad Le Roussillon, Limoges

IPD SHARING:
Plan to Share IPD: No